CLINICAL TRIAL: NCT06886256
Title: Enabling Access to Prehabilitation for Kidney Transplant Candidates Who Are Frail
Brief Title: Prehabilitation for Kidney Transplant Candidates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Atiya Dhala, Associate Professor of Clinical Medicine in Clinical Surgery, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00038084
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplantation; Frailty; Chronic Kidney Insufficiency
Keywords: Kidney Transplantation; Frailty; Chronic Kidney Insufficiency
MeSH Terms: conditions — Frailty; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Each participant will have 3 wearable sensors placed during a single exercise event. The data collected from the sensors will be transferred to a mHealth platform for monitoring feasibility.
  Interventions: Device: Polar H10 Heart Rate Monitor; Device: Empatica EmbracePlus; Device: Apple Watch Ultra 2

INTERVENTIONS:
Device: Polar H10 Heart Rate Monitor — Wearable sensors to capture movement-based data during physical therapy session. The Polar H10 Heart Rate Monitor measures heart rate and will transfer the data to the mHealth app.
Device: Empatica EmbracePlus — Wearable sensors to capture movement-based data during physical therapy session. The Empatica EmbracePlus measures physiological parameters and will transfer the data to the mHealth app.
Device: Apple Watch Ultra 2 — Wearable sensors to capture movement-based data during physical therapy session. The Apple Watch Ultra 2 measures heart rate, will transfer the data to the mHealth app, and will provide an alert when the heart rate is too high or too low.

SUMMARY:
This interventional trial seeks to determine the feasibility of wearable sensors to provide data from patients while undergoing supervised exercise.

DETAILED DESCRIPTION:
This pilot study is a prospective, non-randomized, interventional trial of measures of prehabilitation in kidney transplant candidates who are frail. Kidney transplant candidates who meet criteria for the study will have wearable sensors placed for monitoring during the exercise session of their prehabilitation. The sensors will capture data during the single exercise session and transfer the data to a mobile health (mHealth) platform. The study aims to use the information from the sensors to develop future studies where the exercise is adjusted based on the sensor reports.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Frail patients who are being evaluated for kidney transplant at Houston Methodist Hospital
2. Male or Female, aged 55 or older
3. Provision of signed and dated informed consent by the participant
4. Willingness to comply with study procedures and the duration of the study

Exclusion Criteria:

1. Inability or contraindication to exercise
2. Refusal to participate
3. Inability to consent or effectively communicate

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieve at least 20 minutes of moderate-intensity exercise during a 1-hour physical therapy session at Visit 2 is greater than 75%. | Day 1
  Moderate intensity exercise is defined as a score of 3-5 on the Modified BORG CR10 Rating Perceived Exertion (RPE)

SECONDARY OUTCOMES:
Muscle strength - Grip strength | Baseline
  hand-held dynamometer, Newtons; Measures upper body strength
Muscle strength - Chair stand test | Baseline
  Number of times from chair sitting to standing in 30 seconds; Measures lower body strength and balance
Physical performance - Gait speed | Baseline
  meters per second; Measures walking speed over a short distance
Physical performance - Timed up and go | Baseline
  seconds; time to stand up from a chair, walk a short distance, turn around, walk back to the chair, and sit down; Assess mobility and balance
Physical performance - Walking test, 6-minute walk | Baseline
  6-minute walk distance, meters; If the test is not available a 5-meter test can be used
Physical performance - Walking test, 5-meter walk | Baseline
  5-meter test, seconds; If the 6-minute walk test is not available a 5-meter test can be used
Respiratory capacity - Maximal inspiratory pressure | Baseline
  Record in units of cmH20; Measure of strength of inspiratory muscles
Respiratory capacity - Adjust Inspiratory Muscle Trainer completion | Baseline
  A binary assessment of whether the inspiratory muscle trainer required adjustment
Physical therapy - Aerobic exercise | Day 1
  Rate of perceived exertion as measured by Modified BORG CR10 Rating Perceived Exertion (RPE) scale of 0 (no exertion or resting) to 10 (pushing yourself to the max).
Physical therapy - Resistance exercise | Day 1
  Rate of perceived exertion as measured by Modified BORG CR10 Rating Perceived Exertion (RPE) scale of 0 (no exertion or resting) to 10 (pushing yourself to the max).

CONTACTS AND LOCATIONS:
Overall Officials: Atyia Dhala, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing will be available from this study.

REFERENCES:
- [Background] Lorenz EC, Hickson LJ, Weatherly RM, Thompson KL, Walker HA, Rasmussen JM, Stewart TL, Garrett JK, Amer H, Kennedy CC. Protocolized exercise improves frailty parameters and lower extremity impairment: A promising prehabilitation strategy for kidney transplant candidates. Clin Transplant. 2020 Sep;34(9):e14017. doi: 10.1111/ctr.14017. Epub 2020 Jul 24. PMID 32573816
- [Background] Yamagami M, Mack K, Mankoff J, Steele KM. "I'm Just Overwhelmed": Investigating Physical Therapy Accessibility and Technology Interventions for People with Disabilities and/or Chronic Conditions. ACM Transactions on Accessible Computing. 2022;15(4):1-22. doi: doi.org/10.1145/3563396.